CLINICAL TRIAL: NCT01648101
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multicentre Study to Determine the Efficacy and Safety of 2 Doses of Retigabine Immediate Release (900 mg/Day and 600 mg/Day) Used as Adjunctive Therapy in Adult Asian Subjects With Drug-resistant Partial-onset Seizures.
Brief Title: Assessment of the Efficacy and Safety of 2 Doses of Retigabine Immediate Release (900 mg/Day and 600 mg/Day) Used as Adjunctive Therapy in Adult Asian Subjects With Drug-resistant Partial-onset Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Registration of the medicine is no longer being pursued in South Korea, Taiwan or Vietnam
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114855
Record Dates: First submitted 2012-06-28; First posted 2012-07-24 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
Keywords: Retigabine IR; Asian Subjects; Adjunctive Therapy; Efficacy; Drug-Resistant; Safety & tolerability; Partial-Onset Seizures; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Retigabine 900mg (Experimental): 900mg total daily dose
  Interventions: Drug: Retigabine 900mg/day
- Retigabine 600mg (Experimental): 600mg total daily dose
  Interventions: Drug: Retigabine 600mg/day
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Retigabine 900mg/day — Study drug will be administered three times a day in a double blind manner. The starting dose of retigabine will be 300 mg/day. This dose will be increased by 150 mg/day per week to reach the target dose of 900mg/day over a 4 week Titration Phase). The subject will then continue to receive 900mg/day for the next 12 weeks (Maintenance Phase). Eligible subjects will then be offered an opportunity to enter an open label extension (OLE) study. After a 4 week transition phase, eligible subjects will start the OLE on retigabine 900mg/day.
  Arms: Retigabine 900mg
Drug: Retigabine 600mg/day — Study drug will be administered three times a day in a double blind manner. The starting dose of retigabine will be 300mg/day. This dose will be increased by 150 mg/day per week to reach the target dose of 600mg/day over 2 weeks. The subject will then continue to receive 600mg/day for the next 14 weeks (2 weeks of the Titration Phase and 12 weeks of the Maintenance Phase). Eligible subjects will then be offered an opportunity to enter an open label extension (OLE) study. After a 4 week Transition Phase (3 weeks on retigabine 600mg/day, 1 week on retigabine 750mg/day) eligible subjects will start the OLE on retigabine 900mg/day.
  Arms: Retigabine 600mg
Other: Placebo — Study drug will be administered three times a day in a double blind manner. Subjects randomised to placebo will receive the same number, size and colour of tablets as the 600mg/day and 900mg/day treatment arms for the duration of the 4 week Titration Phase and the 12 week Maintenance Phase. Eligible subjects will then be offered an opportunity to enter an open label extension (OLE) study. The starting dose of retigabine will be 300 mg/day. This dose will be increased by 150 mg/day per week to reach dose of 750mg/day over the 4 weeks of the Transition Phase. On completion of the Transition Phase eligible subjects will start the OLE on retigabine 900mg/day.
  Arms: Placebo

SUMMARY:
The immediate release (IR) formulation of retigabine has been shown to be superior to placebo as adjunctive therapy in 3 adequate and well-controlled studies in subjects with drug-resistant partial-onset seizures (POS) who had previously failed to respond to two or more antiepileptic drugs (AEDs) and were still having seizures despite current treatment with 1, 2, or 3 AEDs. However, of 1244 subjects randomly assigned to treatment in these 3 clinical studies, only 10 were Asian subjects and only 5 of these Asian subjects were randomly assigned to treatment with retigabine. Therefore, this Phase III study is being conducted to evaluate the efficacy, safety and tolerability, and health outcomes of retigabine, at doses of 900 mg/day and 600 mg/day, compared with placebo in adult Asian subjects with drug-resistant POS.

DETAILED DESCRIPTION:
This is a Phase III study evaluating the efficacy, safety and tolerability, and health outcomes of 2 doses of retigabine immediate release (IR) (GW582892) compared with placebo in adult Asian subjects with drug-resistant partial-onset seizures (POS) who are already taking 1, 2, or 3 antiepileptic drugs (AEDs). This randomised, double-blind, placebo-controlled, parallel-group study will compare retigabine IR at doses of 900 mg/day and 600 mg/day taken in equally divided doses three times a day with placebo.

The study design includes an 8-week Screening/Baseline Phase, a 16-week Treatment Phase (4-week Titration Phase and 12-week Maintenance Phase), and a 4-week Transition or Taper/Follow-up Phase. Approximately 500 subjects will be screened and enrolled with approximately 354 subjects randomly assigned to 1 of 3 treatment groups in a ratio of 1:1:1 (retigabine 900 mg/day, retigabine 600 mg/day, or placebo). The total duration of the study for each subject will be approximately 28 weeks. At the end of the Maintenance Phase, eligible subjects will be given the opportunity to enrol in an open-label extension study.

The primary efficacy endpoint is the proportion of responders, defined as subjects with >/=50% reduction in 28 day total POS frequency, from the Baseline Phase to the Maintenance Phase, in subjects randomly assigned to retigabine 900 mg/day compared with placebo. The key secondary efficacy endpoint is the proportion of responders, defined as subjects with >/=50% reduction in 28 day total POS frequency, from the Baseline Phase to the Maintenance Phase, in subjects randomly assigned to retigabine 600 mg/day compared with placebo.

The safety and tolerability endpoints are incidence and severity of adverse events (AEs); proportion of subjects with AEs leading to discontinuation; change from Baseline in vital sign measurements and weight; change from Baseline in electrocardiogram parameters; change from Baseline in haematology, chemistry, and urinalysis parameters; changes from Baseline in American Urological Association Symptom Index and post-void residual bladder ultrasound volumes; and summary of the Columbia-Suicide Severity Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

* Asian men or women ≥18 years of age at the time of consent.
* Have a confident diagnosis of epilepsy with POS with or without secondary generalisation (classified according to International League Against Epilepsy, 1981) for ≥2 years and is having POS despite having been treated in the past with ≥2 approved AEDs either alone or together at adequate doses for a sufficient length of time in the opinion of the investigator.
* Have had, within the last 10 years, 1 electroencephalogram or video electroencephalogram and 1 brain magnetic resonance imaging or computerised tomography scan with results consistent with a diagnosis of POS. If diagnostic studies are negative and if history during clinical assessment suggests a diagnosis of POS, and other diseases have been excluded, the subject can be enrolled.
* Have a documented 28-day partial seizure frequency rate of ≥4 partial seizures over the 8 weeks preceding the screening visit. subjects should not be seizure free for ≥21 consecutive days. In subjects with simple partial seizures, only seizures with motor signs will be counted towards meeting the inclusion criteria.
* Currently being treated with a stable regimen of 1, 2, or 3 AEDs for ≥1 month prior to the screening visit. If the subject is taking barbiturates (e.g., phenobarbital), the dose of the barbiturate must have been stable for ≥3 months prior to the screening visit Note: Vagus Nerve Stimulator: VNS will not be counted as a concurrent AED. Subjects with surgically implanted VNS will be allowed to enter the study provided that all of the following conditions are met: a. The VNS has been in place for ≥6 months prior to the screening visit; b. The settings must have remained constant for ≥1 month prior to the screening visit and remain constant throughout the study; c. The battery is expected to last for the duration of the study; d. Subjects who are considering implantation of a VNS are excluded from participation in the study. Note: Benzodiazepines: The chronic use of a benzodiazepine as a concurrent AED is permitted as long as the dose is kept constant for ≥1 month prior to the screening visit and remains constant throughout the study.
* Able and willing to maintain an accurate and complete daily written seizure calendar or has a caregiver who is able and willing to maintain an accurate and complete daily written seizure calendar.
* Able to understand and willing to provide written informed consent, or has a legally authorised representative able to so, before any protocol-specific procedures are performed.
* A female subject is eligible to enter and participate in the study if she is: a. Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is postmenopausal); Premenopausal females with a documented (medical report verification) hysterectomy with or without oophorectomy or bilateral oophorectomy when reproductive status has been confirmed by hormone level assessment; Postmenopausal females defined as being amenorrheic for greater than 1 year with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms). However, if indicated, this should be confirmed by estradiol and follicle-stimulating hormone levels consistent with menopause (according to local laboratory ranges). Women who have not been confirmed as postmenopausal should be advised to use contraception as listed in the protocol: b. Of childbearing potential, has a negative serum pregnancy test at Screening and a negative urine and serum pregnancy test at randomisation, and agrees to satisfy one of the requirements listed in the protocol: c. Not pregnant or lactating (breastfeeding) or planning to become pregnant during the study.
* Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2 times the upper limit of normal (ULN); alkaline phosphatase (ALP) and bilirubin </=1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Have generalised epilepsy (such as Lennox-Gastaut syndrome, juvenile myoclonic epilepsy, absence epilepsy, etc.), innumerable seizures within the 12-month period prior to study entry where the individual seizures cannot be counted, or nonepileptic seizures.
* Have had status epilepticus (other than simple partial status epilepticus) within the 12 months prior to Screening.
* Have had previous exposure to retigabine.
* Have impaired renal function as judged by a creatinine clearance of <50 mL/min.
* Have a history of substance abuse (alcohol or drugs) or substance dependence within 12 months prior to Screening.
* Have taken an investigational drug, or used an investigational device, within the 30 days prior to Screening or plans to take another investigational drug at any time during the study.
* Are currently following or planning to follow a ketogenic diet.
* Have been treated with felbamate or vigabatrin within the 6 months prior to Screening. If a subject has been previously treated with vigabatrin >6 months prior to Screening, a visual perimetry test performed within 6 months prior to Screening must show normal visual fields or no worsening of recognised visual field abnormalities as compared with prior to vigabatrin treatment.
* Are using central nervous system (CNS)-active medication (other than concomitant AED therapy), unless the subject has been stabilised on such medication for more than 1 month prior to Screening; or currently taking medications known to lower seizure threshold (e.g., antipsychotics) and monoamine oxidase (MAO) inhibitors.
* Are using herbal treatments with CNS activity within 1 month prior to Screening.
* Are planning surgery during the study to control seizures.
* Are suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormalities that are likely to interfere with the objectives of the study.
* Have a history of urinary retention or risk factors for urinary retention that in the investigator's judgment could potentially affect subject safety.
* Have any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to: clinically significant cardiac, renal, or hepatic conditions; or a condition that affects the absorption, distribution, metabolism or excretion of drugs.
* Have an average corrected QT interval (QTc; either QTcB Bazett's correction or QTcF Fridericia's correction) ≥450 msec or ≥480 msec for subjects with bundle branch block at the time of Screening.
* Have active suicidal plan/intent or have had active suicidal thoughts in the past 6 months. Have a history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Have a history of malignancy within the past 2 years, with the exception of basal cell carcinoma.
* Have a known hypersensitivity to any components of the study medication.

Randomisation Criteria:

Subjects must also meet the following criteria at the end of the Baseline Phase (Visit 3) and before randomisation and administration of the first dose of study medication:

* Have a documented 28-day total POS frequency rate of ≥4 POS over an 8 week Baseline Phase. Note: In subjects with simple partial seizures, although all seizures occurring during the Baseline Phase will be collected, only seizures with motor signs will be counted toward qualification for meeting the randomisation criteria.
* Have not had a seizure-free period of ≥21 consecutive days during the Baseline Phase.
* Have not had innumerable seizures (defined as an episode of seizure activity lasting <30 minutes during which several seizures occur with such frequency that the initiation and termination of each individual seizure cannot be distinguished) during the 8 week Baseline Phase.
* Have not had an episode of status epilepticus (other than simple partial status epilepticus) during the 8 week Baseline Phase
* Have not required dose adjustments of concurrent AEDs, addition of new AEDs, discontinuation of existing AEDs, changes to VNS settings, or acute use of benzodiazepines for the treatment of seizures during the Baseline Phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08-29; Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- Hong Kong (4):
  - GSK Investigational Site, Hang Hau
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Shatin
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seberang Jaya
- Philippines (3):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Manila
- GSK Investigational Site, Singapore, Singapore
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Taiwan (8):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiumg
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Proposal for revised clinical and electroencephalographic classification of epileptic seizures. From the Commission on Classification and Terminology of the International League Against Epilepsy. Epilepsia. 1981 Aug;22(4):489-501. doi: 10.1111/j.1528-1157.1981.tb06159.x. No abstract available. PMID 6790275
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114855 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with drug-resistant partial-onset seizures (POS) who were taking 1, 2, or 3 antiepileptic drugs (AEDs) with or without vagus nerve stimulator (VNS); had a 28-day total POS frequency rate >=4 seizures; and did not have a period of >=21 consecutive days without a POS over the 8-week Baseline Phase were enrolled in this study.
Pre-assignment Details: 76 participants (par.) were randomized to study treatment; 75 par. comprised the Intent-to-Treat Population (par. who were randomly assigned to treatment, received >=1 dose/any portion of a dose of study medication, had Baseline [BL] seizure data, and had >=1 post-BL seizure record between the Titration Phase and the end of the Maintenance Phase).
Groups:
- Placebo: Participants entered a 16-week Treatment Phase (TrP) consisting of a 4-week Titration Phase (TiP) and a 12-week Maintenance Phase (MP). In the TiP, participants received matching placebo in increasing doses. Participants that could not tolerate the titration or withdrew were discontinued from the study and entered the Taper/Follow-up Phase (TaP/FUP). Participants who tolerated titration entered the MP and continued to receive the same dose regimen for 12 weeks. After completing the MP, participants who opted to enroll in the open-label extension (OLE) study entered the 4-week Transition Phase (TnP). In the TnP, participants received active retigabine in increasing doses starting at 300 milligrams per day (mg/day), 450 mg/day, 600 mg/day, and 750 mg/day, respectively, in each of 4 weeks. Participants that did not enroll in the OLE study completed a 3-week TaP and 1 week of FUP.
- Retigabine 600 mg/Day: Participants entered a 16-week TrP consisting of a 4-week TiP and a 12-week MP. In the TiP, participants received a starting dose of retigabine (RTG) 300 mg/day that increased by 150 mg/day per week until a target dose of 600 mg/day was reached. Participants that could not tolerate the titration or withdrew were discontinued from the study and entered the TaP/FUP. Participants who tolerated titration entered the MP and continued to receive 600 mg/day for 12 weeks. After completing the MP, participants who opted to enroll in the OLE study entered the 4-week TnP. In the TnP, participants received RTG 600 mg/day for 3 weeks and RTG 750 mg/day in the last week. Participants that did not enroll in the OLE study completed a 3-week TaP and 1 week of FUP.
- Retigabine 900 mg/Day: Participants entered a 16-week TrP consisting of a 4-week TiP and a 12-week MP. In the TiP, participants received a starting dose of RTG 300 mg/day that increased by 150 mg/day per week until a target dose of 900 mg/day was reached. Participants that could not tolerate the titration or withdrew were discontinued from the study and entered the TaP/FUP. Participants who tolerated titration entered the MP and continued to receive 900 mg/day for 12 weeks. After completing the MP, participants who opted to enroll in the OLE study entered the 4-week TnP. In the TnP, participants received RTG 900 mg/day for 4 weeks. Participants that did not enroll in the OLE study completed a 3-week TaP and 1 week of FUP.
Period: Titration Phase (4 Weeks)
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Started | 25 | 26 | 24
Completed | 23 | 23 | 18
Not Completed | 2 | 3 | 6
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Reached Protocol Defined Criteria | 0 | 0 | 1
Period: Maintenance Phase (12 Weeks)
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Started | 23 | 23 | 18
Completed | 20 | 20 | 12
Not Completed | 3 | 3 | 6
Not completed — Withdrew Consent | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Adverse Event | 1 | 3 | 4
Period: Transition Phase (4 Weeks)
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Started | 17 (After completing the MP, only those par. that chose to enter the OLE study started the TnP) | 18 (After completing the MP, only those par. that chose to enter the OLE study started the TnP) | 9 (After completing the MP, only those par. that chose to enter the OLE study started the TnP)
Completed | 12 | 13 | 5
Not Completed | 5 | 5 | 4
Not completed — Adverse Event | 4 | 3 | 2
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Study Terminated | 1 | 0 | 0
Period: Taper/Follow-up Phase (4 Weeks)
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Started | 1 (Includes only those par. who completed the Titration + MN phase, but opted not to enroll in the OLE) | 2 (Includes only those par. who completed the Titration + MN phase, but opted not to enroll in the OLE) | 3 (Includes only those par. who completed the Titration + MN phase, but opted not to enroll in the OLE)
Completed | 1 | 1 | 3
Not Completed | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retigabine 900 mg/Day | Retigabine 600 mg/Day | Placebo | Total
Number analyzed (Participants) | 24 | 26 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for members of the Safety Population: all randomized participants who received at least one dose of study medication.
  Years | 36.0 (9.43) | 37.1 (10.90) | 36.3 (13.50) | 36.5 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data are reported for members of the Safety Population: all randomized participants who received at least one dose of study medication.
  Participants
    Female | 10 | 10 | 10 | 30
    Male | 14 | 16 | 15 | 45
Race/Ethnicity, Customized [Number; unit: Participants] — Baseline data are reported for members of the Safety Population: all randomized participants who received at least one dose of study medication.
  Participants
    Asian - East Asian Heritage | 17 | 16 | 15 | 48
    Asian - South East Asian Heritage | 7 | 10 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Placebo and Retigabine 900 mg Responders During the Maintenance Phase (MP)
Description: A responder is defined as a par. with >=50% reduction in the 28 day total partial on-set seizure (POS) frequency from the Baseline Phase (BP) to the MP, randomly assigned to retigabine 900 mg/day compared with placebo. The total 28-day POS rate was defined as: (total number of POS over the evaluable period (MP) / number of days of seizure (sz) data in the evaluable period) *28 days. In the event of one or more innumerable seizures (IS) occurring on a day, these were to be counted as an additional 10 seizures for that day, regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of MP minus start date of the MP minus days on which seizures were recorded as "Not done" + 1). Each occurrence of status epilepticus (SE) was counted as 1 seizure (whether partial or not).
Time Frame: Baseline (BL); Week 4 up to Week 16
Population: ITT Population: all par. who were randomly assigned to treatment; rec'd≥1 dose (or any portion of dose) of study medication; had BL sz data; and had ≥1 post-BL sz record (whether or not they had a sz) between start of TiP and end of MP. Par. who dropped out during TiP were classified as non-responders. For all other par. only MP data were used.
Measure: Number; unit: Participants
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 0 | 24
Participants
  Responders | 0 |  | 4
  Non-Responders | 25 |  | 20

2. Secondary Outcome: Number of Placebo and Retigabine 600 mg Responders During the MP
Description: A "responder" is defined as a participant experiencing a >=50% reduction in the 28-day total POS frequency from the BP to the MP, randomly assigned to retigabine 600 mg/day compared to placebo. The 28-day total POS frequency was calculated as: (total number of PS over the time period of interest [MP] / number of applicable days in that period) * 28. In a case of one or more occurrences of IS on a day, these seizures were to be counted as an additional 10 seizures for that day, regardless of whether the IS were PS or not, and regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of the MP minus the start date of the MP minus days on which seizures were recorded as "Not Done" during the MP plus 1). Each occurrence of SE was counted as 1 seizure (whether partial status or not).
Time Frame: Baseline; Week 4 up to Week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 0
Participants
  Responders | 0 | 8 |
  Non-Responders | 25 | 18 |

3. Secondary Outcome: Number of Responders From the BP to the Treatment Phase (TrP)
Description: A "responder" is defined as a participant experiencing a >=50% reduction in the 28-day total POS frequency from the BP to the TrP (TiP plus MP). The 28-day total POS frequency was calculated as: (total number of PS over the time period of interest [TrP] / number of applicable days in that period) * 28. In a case of one or more occurrences of IS on a day, these seizures were to be counted as an additional 10 seizures for that day, regardless of whether the IS were PS or not, and regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of the TrP minus the start date of the TrP minus days on which seizures were recorded as "Not Done" during the TrP plus 1). Each occurrence of SE was counted as 1 seizure (whether partial status or not).
Time Frame: From Baseline up to Week 16
Population: Intent-to-Treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Participants
  Responders | 1 | 8 | 6
  Non-Responders | 24 | 18 | 18

4. Secondary Outcome: Percent Change From Baseline in the 28-day Total POS Frequency During the MP
Description: The 28-day total POS frequency was calculated as: (total number of PS over the time period of interest [MP] / number of applicable days in that period) * 28. In a case of one or more occurrences of IS on a day, these seizures were to be counted as an additional 10 seizures for that day, regardless of whether the IS were PS or not, and regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of the MP minus the start date of the MP minus days on which seizures were recorded as "Not Done" during the MP plus 1. Percent change from Baseline was calculated as: ([the 28-day PS rate for the period of interest (MP) minus the Baseline 28-day PS rate] / Baseline 28-day PS rate) * 100. A negative percent change indicates a reduction (improvement) from Baseline; thus, the best possible outcome is -100% (100% reduction). There was no theoretical upper limit for worsening.
Time Frame: Baseline; Week 4 up to Week 16
Population: ITT Population. Participants who dropped out during the TiP were calculated based on TiP data. For all others, only MP data were used.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Percent change | -22.21 [-48.6 to 61.0] | -33.90 [-100.0 to 16.3] | -22.46 [-100.0 to 263.63]

5. Secondary Outcome: Percent Change From Baseline in the 28-day Total POS Frequency During the TrP
Description: The 28-day total POS frequency was calculated as: (total number of PS over the time period of interest [TrP; TiP plus MP] / number of applicable days in that period) * 28. In a case of one or more occurrences of IS on a day, these seizures were to be counted as an additional 10 seizures for that day, regardless of whether the IS were PS or not, and regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of the TrP minus the start date of the TrP minus days on which seizures were recorded as "Not Done" during the TrP plus 1. Percent change from Baseline was calculated as: ([the 28-day PS rate for the period of interest (TrP) minus the Baseline 28-day PS rate] / Baseline 28-day PS rate) * 100. A negative percent change indicates a reduction (improvement) from Baseline; thus, the best possible outcome is -100% (100% reduction). There was no theoretical upper limit for worsening.
Time Frame: From Baseline up to Week 16
Population: ITT Population. Participants who dropped out during the TiP were calculated based on TiP data. For all others both Titration and Maintenance Phase data were used
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Percent change | -22.55 [-70.5 to 54.8] | -36.30 [-100.0 to 8.2] | -26.73 [-100.0 to 176.4]

6. Secondary Outcome: Percent Change From Baseline in the 28-day Total POS Frequency During the MP Categorized as: no Change/Increase, >0% to <50% Decrease, 50% to 75% Decrease, and >75% to 100% Decrease
Description: The 28-day total POS frequency was calculated as: (total number of PS over the time period of interest [MP] / number of applicable days in that period) * 28. In a case of >=1 occurrence of IS on a day, these seizures were to be counted as an additional 10 seizures for that day, regardless of whether the IS were PS or not, and regardless of the number of occurrences of IS on that day. The number of applicable days in a phase for seizure data is calculated as: the end date of the MP minus the start date of the MP minus days on which seizures were recorded as "Not Done" during the MP plus 1. Percent change from Baseline was calculated as: ([the 28-day PS rate for the period of interest (MP) minus the Baseline 28-day PS rate] / Baseline 28-day PS rate) * 100. A negative percent change indicates a reduction (improvement) from Baseline. There was no theoretical upper limit for worsening. Each occurrence of status epilepticus (SE) was counted as 1 seizure (whether partial status or not).
Time Frame: Baseline; Week 4 up to Week 16
Population: ITT Population: Due to the early termination of the study, insufficient data are available to perform these analysis.
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in 28 Day Total POS Frequency During the TrP Categorized as: no Change/Increase, >0% to <50% Decrease, 50% to 75% Decrease, and >75% to 100% Decrease
Description: as for outcome 5
Time Frame: From Baseline up to Week 16
Population: ITT Population: Due to the early termination of the study, insufficient data are available to perform these analysis.
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in the 28-day Total POS Frequency During the MP Categorized as: >25% Increase and 0% to 25% Increase
Description: as for outcome 4
Time Frame: Baseline; Week 4 up to Week 16
Population: ITT Population: Due to the early termination of the study, insufficient data are available to perform these analysis.
Arm/Group | Overall Study Arm | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Percent Change From Baseline in the 28-day Total POS Frequency During the TrP Categorized as: >25% Increase and 0% to 25% Increase
Description: as for outcome 5
Time Frame: From Baseline up to Week 16
Population: ITT Population: Due to the early termination of the study, insufficient data are available to perform these analysis.
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Were Seizure Free During the MP, ITT Population
Description: A seizure free-day is defined as a day with non-missing seizure data but without any seizures. A participant was considered to be seizure free during the MP if he/she had no record of countable seizures of any type, no IS, and no SE during the MP. Participants who had one or more days on which they recorded seizures as "Not Done" on the seizure calendar were not disqualified from being considered as seizure free for that day. Participants who did not complete the study or experienced any seizures in the MP were not considered to be seizure free. A participant who completed the study AND had no seizures during the maintenance phase were counted to be seizure free. Also, a completer who only had seizures during the TiP is considered seizure free.
Time Frame: Baseline; Week 4 up to Week 16
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Who Were Seizure Free During the TrP
Description: A seizure free-day is defined as a day with non-missing seizure data but without any seizures. A participant was considered to be seizure free during the TrP if he/she had no record of countable seizures of any type, no IS, and no SE during the TrP. Participants who had one or more days on which they recorded seizures as "Not Done" on the seizure calendar were not disqualified from being considered as seizure free for that day. A participant was considered to be seizure free if they experienced no seizures in the TiP or MP regardless of how long they were in the study.
Time Frame: From Baseline up to Week 16
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Participants | 0 | 1 | 2

12. Secondary Outcome: Percentage of Seizure-free Days in the MP
Description: The percentage of seizure-free days was calculated as: (total number of days without seizures in the MP / number of applicable days in the MP) * 100. A seizure-free day is defined as a day with non-missing seizure data but without any seizures. A participant was considered to be seizure free during the MP if he/she had no record of countable seizures of any type, no IS, and no SE during the MP. Participants who had one or more days on which they recorded seizures as "Not Done" on the seizure calendar were not disqualified from being considered as seizure free for that day.
Time Frame: From Week 4 up to Week 16
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of seizure-free days
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Percentage of seizure-free days | 61.7 (28.31) | 70.6 (31.55) | 63.3 (28.45)

13. Secondary Outcome: Percentage of Seizure-free Days in the TrP
Description: The percentage of seizure-free days was calculated as: (total number of days without seizures in the TrP (TiP plus MP) / number of applicable days in the TrP) * 100. A seizure-free day is defined as a day with non-missing seizure data but without any seizures. A participant was considered to be seizure free during the TrP if he/she had no record of countable seizures of any type, no IS, and no SE during the TrP. Participants who had one or more days on which they recorded seizures as "Not Done" on the seizure calendar were not disqualified from being considered as seizure free for that day.
Time Frame: From Baseline up to Week 16
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of seizure-free days
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Percentage of seizure-free days | 62.1 (27.85) | 70.4 (31.42) | 64.9 (27.47)

14. Secondary Outcome: Incidence of New Seizure Types During the TrP in Participants Without a History of the Indicated Seizure Types at Baseline
Description: A participant was considered to have new seizure types during the TrP if they experienced a new seizure types (such as SE, myoclonic, absence, secondary generalization) and had no prior history of these seizure types. At Screening, a history of previous seizure types was collected, with "Yes," "No," "IS," "SE," or "Unknown" being recorded for each of the seizures types. The history of seizure types was updated during the 8-week BP as pre-treatment status. New types of seizures during the TrP were recorded as A1=simple PS with motor signs; AX=simple PS without motor signs; B=complex PS; C=PS evolving to secondary generalized seizures; D1=absence of seizures; D2=myoclonic seizures; D3=clonic seizures; D4=tonic seizures; D5=tonic-clonic seizures; D6=atonic seizures; E=unclassified seizures; and SE=status epilepticus.
Time Frame: From Baseline up to Week 16
Population: ITT Population.
Measure: Number; unit: Number of events
Arm/Group | Placebo | Retigabine 600 mg/Day | Retigabine 900 mg/Day
Number analyzed (Participants) | 25 | 26 | 24
Number of events
  Simple partial seizures (sz)with motor signs | 2 | 0 | 0
  Partial sz evolving to secondary generalized sz | 0 | 0 | 2
  Complex partial seizures | 0 | 1 | 0
  Simple partial seizures without motor signs | 0 | 0 | 0
  Absence seizures | 0 | 0 | 0
  Myoclonic seizures | 0 | 0 | 0
  Clonic seizures | 0 | 0 | 0
  Tonic seizures | 0 | 0 | 0
  Tonic-clonic seizures | 0 | 0 | 0
  Atonic seizures | 0 | 0 | 0
  Unclassified seizures | 0 | 0 | 0
  Status Epilepticus | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent SAEs and non-serious AEs were collected from start of study treatment until the end of the TnP for participants who entered the OLE study (up to Week 20), or until the follow-up visit for par. who entered the TaP (up to Week 20).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | Retigabine 900 mg/Day | Retigabine 600 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/26 | 1/25
Other Adverse Events (participants affected / at risk) | 20/24 | 24/26 | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retigabine 900 mg/Day (N=24) | Retigabine 600 mg/Day (N=26) | Placebo (N=25)
Dizziness (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retigabine 900 mg/Day (N=24) | Retigabine 600 mg/Day (N=26) | Placebo (N=25)
Dizziness (Nervous system disorders) | 8 | 10 | 6
Somnolence (Nervous system disorders) | 6 | 10 | 4
Tremor (Nervous system disorders) | 2 | 5 | 1
Memory impairment (Nervous system disorders) | 2 | 1 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 5 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Bradyphrenia (Psychiatric disorders) | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
RTG114855 was designed for registration of retigabine as add-on treatment of drug-resistant POS in South Korea/Taiwan/ Vietnam. GSK decided not to pursue registration in these countries and terminated the study early based on new safety information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.